CLINICAL TRIAL: NCT06877689
Title: Expanded Access Protocol of Apitegromab for Patients With Spinal Muscular Atrophy
Brief Title: EAP of Apitegromab for Patients With Spinal Muscular Atrophy
Status: Available | Type: Expanded Access
Sponsor: Scholar Rock, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SRK-015-008
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: SMA
Keywords: Expanded Access; Pre-Approval Access; Compassionate Use
MeSH Terms: interventions — apitegromab

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Apitegromab — Apitegromab (SRK-015) is a fully human anti-proMyostatin monoclonal antibody (mAb) that specifically binds to human pro/latent myostatin, inhibiting myostatin activation. Apitegromab will be administered every 4 weeks by intravenous (IV) infusion.
  Other Names: SRK-015

SUMMARY:
The purpose of this expanded access program (EAP) is to provide access to apitegromab for eligible patients with spinal muscular atrophy (SMA) prior to approval by the local regulatory agency . A medical doctor must decide whether the potential benefit outweighs the risk of receiving an investigational therapy based on the individual patient's medical history and program eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

1. ≥2 years of age.
2. Documented diagnosis of 5q SMA.

Exclusion Criteria:

1. Previous history of a hypersensitivity reaction to a monoclonal antibody or recombinant protein bearing an Fc domain (eg, a soluble receptor-Fc fusion protein), apitegromab, or excipients of apitegromab.
2. Enrolled in a clinical study for any investigational drug.
3. Pregnant or breastfeeding.

Min Age: 2 Years | Sex: All
Age Groups: Child, Adult, Older Adult